CLINICAL TRIAL: NCT06157710
Title: Randomised Controlled Trial of a Digital Programme for Procrastination in UK University Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Collaborators: Uppsala University (Other); Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Jeffrey Lambert, Dr Jeffrey Lambert, University of Bath
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Procrastinate2023
Record Dates: First submitted 2023-11-27; First posted 2023-12-06 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Procrastination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Procrastinate digital programme (Experimental): 8-week unternet-based CBT for procrastination
  * Behavioural Module: Introduction
  * Behavioural Module: Goal setting techniques
  * Behavioural Module: Motivation
  * Behavioural Module: Barriers to action
  * Behavioural Module: Managing maladaptive thoughts and beliefs
  * Behavioural Module: Value clarification
  * Behavioural Module: Moving forward
  Interventions: Behavioral: Digital intervention through modules
- Waitlist control (No Intervention): Wait-list control group. They do not receive the weekly modules though they are asked to complete 4-week and 8-week online surveys.
  They will be allowed to revive the intervention after 8 weeks.

INTERVENTIONS:
Behavioral: Digital intervention through modules — * Introduction
  * Goal Setting Techniques
  * Motivation
  * Barriers to Action
  * Managing Maladaptive Thoughts and Beliefs
  * Value Clarification
  * Moving Forward
  Arms: Procrastinate digital programme

SUMMARY:
The aim of this study is to evaluate the effect of an 8-week self-directed internet based CBT intervention on various psychological outcomes for young students struggling with procrastination in the UK. The psychological outcomes consist of motivation, depressive symptoms, impulsivity and anxiety. More specifically, the study aims to compare the effect of the intervention vs waitlist control at 8 weeks on primary and secondary outcomes. Additionally, the study aims to explore whether changes in primary and secondary outcomes as the result of the intervention are mediated or moderated by key intervention processes.

ELIGIBILITY:
Inclusion Criteria:

* Resident in the UK
* Fluent in English
* Aged between 16 and 24 years of age
* Have access to computer or smartphone
* Score at least 40 points on the Pure Procrastination Scale (indicating difficulties with procrastination)

Exclusion Criteria:

* Ongoing psychological treatment
* New course of change in dose of psychotropic medication in the last two months (self-reported)

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Procrastination: Pure Procrastination Scale (PPS; Rozental, Forsell, et al., 2014) | Baseline, WK4, WK8
  measures procrastination by using 12 items to detect and determine dysfunctional delay. The higher the score the more likely the individual is to delay an activity or task

SECONDARY OUTCOMES:
Demographics | Baseline
  Age, gender, ethnicity, whether they were the first person in their family to attend university, international student status, course type, year of study, and method of recruitment.
Clinical Perfectionism Questionnaire (CPQ) (Fairburn et al., 2003) | Baseline, WK4, WK8
  Assessment of cognitive, behavioural, and affective aspects of setting goals and striving to meet them. This scale has 12 items that assess clinical perfectionism. Items 2 and 8 are reverse-scored.The CPQ items are scored based on the individual's experiences over the past 28 days. The scale utilises a 4-point Likert scale ranging from 1 with the statement "not at all" to 4 with the statement "all the time". Higher scores on the CPQ indicate higher levels of perfectionism.
Depressive symptoms: Patient health questionnaire-8 (PHQ-8) (Kroenke et al., 2008) | Baseline, WK4, WK8
  This assessment measures depressive symptoms. The questionnaire asks how often participants have been bothered or felt affected by eight possible issues or symptoms over the past 2 weeks (e.g., "feeling down, depressed, or hopeless,". The scale consists of eight of the nine criteria to determine depression. A score on the PHQ-8 ≥10 represents clinically significant depression.
Anxiety symptoms: General Anxiety Disorder Scale (GAD-7) (Spitzer et al., 2006) | Baseline, WK4, WK8
  This scale is used to assess anxiety using 7 items relating to worry symptoms in the last 2 weeks. The scores on the scale range from 0 to 21. There are cut off points to indicate different anxiety levels. The scores of 5,10 and 15 show the thresholds for mild anxiety, moderate anxiety, and severe anxiety. participants have been bothered or felt affected by eight possible issues or symptoms over the past 2 weeks (e.g., "feeling down, depressed, or hopeless,". The scale consists of eight of the nine criteria to determine depression. A score on the PHQ-8 ≥10 represents clinically significant depression.
Impulsivity: Short form Barratt Impulsiveness Scale (Spinella 2009) | Baseline, WK4, WK8
  Assessment of 15 items for impulsivity. The scale focuses on non planning, motor impulsivity, and attention impulsivity. Higher scores are indicative of more impulsivity.
International physical activity questionnaire short form (Lee et al., 2011 | Baseline, WK4, WK8
  The questionnaire consists of 9 items and it asks participants about their physical activity in the last 7 days before completing the form. It explores how often participants engaged with physical activity ranging at four levels: vigorous-intensity, moderate-intensity, walking, and sitting.
Behavioural activation for depression scale (BATDS-SF) (Manos et al., 2011) | Baseline, WK4, WK8
  Assessment of experienced pleasure from daily activities over the past week. It consists of 9 items on 7 point scales from 0 to 6. 0 being "not at all" to 6 "completely".
Intervention acceptability and appropriateness using the Intervention Appropriateness Measure (IAM), acceptability of Interventions Measure (AIM) and feasibility of intervention measure | WK4, WK8
  This scale is used to measure how appropriate the intervention will be on the participants. This assessment uses 4 item measures which focus on how likely it is that the implementation of the intervention will be successful on the participants.
Usage data from intervention platform (e.g., time spend on modules, completion of worksheets) | Baseline to WK8
  Assessing how far and how much of each module was completed based on time spent and whether worksheets were completed.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bath, Bath, United Kingdom

IPD SHARING:
Plan to Share IPD: No